CLINICAL TRIAL: NCT04517994
Title: Strength at Home Couples Program to Prevent Military Partner Violence
Brief Title: Implementation of Strength at Home for Military Couples
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston VA Research Institute, Inc. (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Casey Taft, Psychologist, Behavioral Sciences Division, National Center for PTSD; Assoc. Professor of Psychiatry, VA Boston Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CDMRP-PT140092
Record Dates: First submitted 2018-01-26; First posted 2020-08-19 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Intimate Partner Violence
Keywords: Prevention; Domestic Violence; Military Couples; Veterans; Marital Relationship; Trauma; PTSD; Implementation
MeSH Terms: conditions — Wounds and Injuries; Stress Disorders, Post-Traumatic | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Treatment (Experimental): The intervention includes components from empirically validated interventions for intimate relationship difficulties and PTSD. This includes core themes of trust, self-esteem, power and control, conflict-management skills, and communication skills training.
  Interventions: Behavioral: Active Treatment
- Supportive Treatment (Active Comparator): Broadly based on the principles and techniques of client centered (Rogerian) therapy, and the fundamental principles and practices for experiential group psychotherapy as specified by Yalom. The group also draws upon the work of Murphy's Supportive Therapy protocol specifically for group intervention with domestic abuse perpetrators.
  Interventions: Behavioral: Supportive Treatment

INTERVENTIONS:
Behavioral: Active Treatment — See arm description.
  Arms: Active Treatment
Behavioral: Supportive Treatment — See arm description.
  Arms: Supportive Treatment

SUMMARY:
The Strength at Home Couples program is designed to enhance intimate relationships and prevent intimate partner violence (IPV) among service members and their partners in light of the unique stressors and experiences of this population.

DETAILED DESCRIPTION:
A Hybrid Type-I Implementation-effectiveness research design will allow the research team, comprising investigators with expertise in treatment development, efficacy and effectiveness research, and implementation science, to simultaneously investigate the effectiveness of SAH-C in a military population while identifying any barriers to implementation that would need to be addressed before SAH-C could be successfully implemented on a larger scale.

SAH-C derives from a unique fusion of interventions for trauma and IPA, integrating elements of cognitive processing therapy for PTSD,39 couples therapy for PTSD,40 and a cognitive behavioral intervention for IPA.41 SAH-C consists of 10 two-hour weekly sessions, co-led by two therapists. This was the minimum length deemed necessary to incorporate components addressing the proposed IPA mechanisms and is consistent with the briefest IPA interventions.42 During each session, couples are provided assignments to practice skills together and to assist with the consolidation of material. A group couples format is used because group cohesion among clients appears to be associated with IPA prevention.43 Group interventions also use less time and resources than individual-based interventions.

ELIGIBILITY:
Inclusion Criteria:

* Couples must be in an intimate relationship
* Must be over the age of 18
* Both members of the couple report no occurrence of physical IPA in the past 3 months and no severe aggression in the past 12
* At least one member reports at or below a score of 100 on the Dyadic Adjustment Scale
* Both members must provide research consent

Exclusion Criteria:

* Will be excluded on the basis of reading difficulties that preclude valid completion of the assessment instruments

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Domestic Violence Prevention - Revised Conflict Tactics Scale (CTS2) | Intake/Pre-Treatment
  Changes of physical and psychological IPV as evidenced by change in CTS2 responses. Each item response option ranges in value from 0-7 with 0 being the minimum value and 7 being the maximum value. Scale is a 78-item measure with higher scores meaning greater conflict.
Domestic Violence Prevention - Change in CTS2 | Post-treatment (after 10 weeks of class)
  Changes of physical and psychological IPV as evidenced by change in CTS2 responses. Each item response option ranges in value from 0-7 with 0 being the minimum value and 7 being the maximum value. Scale is a 78-item measure with higher scores meaning greater conflict.
Domestic Violence Prevention - Change in CTS2 | 3-month post-group follow-up (3-months after last class)
  Changes of physical and psychological IPV as evidenced by change in CTS2 responses. Each item response option ranges in value from 0-7 with 0 being the minimum value and 7 being the maximum value. Scale is a 78-item measure with higher scores meaning greater conflict.
Relationship Satisfaction: Dyadic Adjustment Scale | Intake/Pre-Treatment
  Changes in relationship satisfaction as evidenced by answers to the Dyadic Adjustment Scale. Items 1-15 options: Always Agree, Almost Always Agree, Occasionally Disagree, Frequently Disagree, Almost Always Disagree, Always Disagree. Item 16-22: All the Time, Most of the Time, More Often than Not, Rarely, Never. Item 23: Every day, Almost Every Day, Occasionally, Rarely, Never. Item 24: All of them, Most of them, Some of them, Very few of them, None of them. Items 25-28: Never, Less than once a month, Once or twice a month, Once or twice a week, Once a day, More often. Items 29-30: Yes/No. Item 31: Extremely Unhappy, Fairly Unhappy, A Little Unhappy, Happy, Very Happy, Extremely Happy, Perfect. Item 32: six statements in which the participant picks the statement that best describes how they feel about the future of their relationship. Overall score ranges from 0 to 151; higher scores indicating a more positive adjustment and lower level of distress within relationship.
Change in Relationship Satisfaction: Dyadic Adjustment Scale | Post-treatment (after 10 weeks of class)
  Changes in relationship satisfaction as evidenced by answers to the Dyadic Adjustment Scale. Items 1-15 options: Always Agree, Almost Always Agree, Occasionally Disagree, Frequently Disagree, Almost Always Disagree, Always Disagree. Item 16-22: All the Time, Most of the Time, More Often than Not, Rarely, Never. Item 23: Every day, Almost Every Day, Occasionally, Rarely, Never. Item 24: All of them, Most of them, Some of them, Very few of them, None of them. Items 25-28: Never, Less than once a month, Once or twice a month, Once or twice a week, Once a day, More often. Items 29-30: Yes/No. Item 31: Extremely Unhappy, Fairly Unhappy, A Little Unhappy, Happy, Very Happy, Extremely Happy, Perfect. Item 32: six statements in which the participant picks the statement that best describes how they feel about the future of their relationship. Overall score ranges from 0 to 151; higher scores indicating a more positive adjustment and lower level of distress within relationship.
Change in Relationship Satisfaction: Dyadic Adjustment Scale | 3-month post-group follow-up (3-months after last class)
  Changes in relationship satisfaction as evidenced by answers to the Dyadic Adjustment Scale. Items 1-15 options: Always Agree, Almost Always Agree, Occasionally Disagree, Frequently Disagree, Almost Always Disagree, Always Disagree. Item 16-22: All the Time, Most of the Time, More Often than Not, Rarely, Never. Item 23: Every day, Almost Every Day, Occasionally, Rarely, Never. Item 24: All of them, Most of them, Some of them, Very few of them, None of them. Items 25-28: Never, Less than once a month, Once or twice a month, Once or twice a week, Once a day, More often. Items 29-30: Yes/No. Item 31: Extremely Unhappy, Fairly Unhappy, A Little Unhappy, Happy, Very Happy, Extremely Happy, Perfect. Item 32: six statements in which the participant picks the statement that best describes how they feel about the future of their relationship. Overall score ranges from 0 to 151; higher scores indicating a more positive adjustment and lower level of distress within relationship.
Domestic Violence Prevention - Multidimensional Measure of Emotional Abuse (MMEA) | Intake/Pre-Treatment
  Changes of physical and psychological IPV as evidenced by changes in MMEA scores. MMEA is a 28-item measurement tool with scale responses ranging from 0 to 7 where higher scores indicate greater emotional abuse.
Domestic Violence Prevention - Change in MMEA | Post-treatment (after 10 weeks of class)
  Changes of physical and psychological IPV as evidenced by changes in MMEA scores. MMEA is a 28-item measurement tool with scale responses ranging from 0 to 7 where higher scores indicate greater emotional abuse.
Domestic Violence Prevention - Change in MMEA | 3-month post-group follow-up (3-months after last class)
  Changes of physical and psychological IPV as evidenced by changes in MMEA scores. MMEA is a 28-item measurement tool with scale responses ranging from 0 to 7 where higher scores indicate greater emotional abuse.

SECONDARY OUTCOMES:
Suicidal Ideation | Intake/Pre-Treatment
  Changes in suicidal ideation through the suicidality measure asking about suicidal thoughts (the four response options include: I do not have thoughts, Sometimes I have thoughts, Most of the time I have thoughts, and I always have thoughts), suicide attempts (response is a fill in the blank), wish to live/die (the three response options include I have a moderate to strong wish to live/die, I have a weak wish to live/die, and I have no wish to live/die), and belongingness (some items will be reverse scored and the 7-point Likert scale includes 1[Not at all true for me], 2, 3, 4 [Somewhat true for me], 5, 6, 7 [Very true for me]). Lower scores indicate less suicidal ideation.
Suicidal Ideation | Post-treatment (after 10 weeks of class)
  Changes in suicidal ideation through the suicidality measure asking about suicidal thoughts (the four response options include: I do not have thoughts, Sometimes I have thoughts, Most of the time I have thoughts, and I always have thoughts), suicide attempts (response is a fill in the blank), wish to live/die (the three response options include I have a moderate to strong wish to live/die, I have a weak wish to live/die, and I have no wish to live/die), and belongingness (some items will be reverse scored and the 7-point Likert scale includes 1[Not at all true for me], 2, 3, 4 [Somewhat true for me], 5, 6, 7 [Very true for me]). Lower scores indicate less suicidal ideation.
Suicidal Ideation | 3-month post-group follow-up (3-months after last class)
  Changes in suicidal ideation through the suicidality measure asking about suicidal thoughts (the four response options include: I do not have thoughts, Sometimes I have thoughts, Most of the time I have thoughts, and I always have thoughts), suicide attempts (response is a fill in the blank), wish to live/die (the three response options include I have a moderate to strong wish to live/die, I have a weak wish to live/die, and I have no wish to live/die), and belongingness (some items will be reverse scored and the 7-point Likert scale includes 1[Not at all true for me], 2, 3, 4 [Somewhat true for me], 5, 6, 7 [Very true for me]). Lower scores indicate less suicidal ideation.

CONTACTS AND LOCATIONS:
Locations (1):
- Joint Base Lewis McChord, Tacoma, Washington, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-15): https://cdn.clinicaltrials.gov/large-docs/94/NCT04517994/Prot_SAP_000.pdf